CLINICAL TRIAL: NCT03585218
Title: Clinical, Emotional, Cognitive and Neuropsychophysiological Impact of a Hedonic Aroma in Women With Breast Cancer Undergoing Chemotherapy: Implications in Quality of Life.
Brief Title: Women With Breast Cancer Undergoing Chemotherapy: Implications in Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minho (Other)
Collaborators: Foundation for Science and Technology, Portugal (Other)
Responsible Party: Principal Investigator, Marta Alexandra Marques Pereira, Principal Investigator, University of Minho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 175519021995
Record Dates: First submitted 2018-05-28; First posted 2018-07-12 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Breast Cancer Female
Keywords: Quality of Life; Breast Cancer; Essentials Oils; Adjuvant Chemotherapy; Salivary cortisol; Neuropsychophysiology
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: On each moment of data collection, the researcher will apply the evaluation protocol to the participant regardless of the group and before chemotherapy treatment. Regarding the psychophysiological variable, each participant's saliva will be collected using salivettes®, while cortisol concentrations will be analyzed through ELISA kits. At the time of the sample collection, before the CT, the participant who accepted to participate and fulfilled the inclusion criteria will be provided with three salivettes and an explanatory leaflet so that, on the day before the 2nd Cycle, they can collect their own saliva, around 23h, and on the day of CT, on waking up and thirty minutes after, fasting. This process will be replicated throughout the remaining evaluation moments. Subsequently, it is also our goal to evaluate the cortisol levels to CT by performing one collection of saliva before and another thirty minutes after CT.
Who Masked: Participant
Masking Description: When a participant is eligible, according to the inclusion criteria, she is allocated to one of the groups in a 1:1 ratio. The randomization assignment was placed in sealed envelopes and assigned before chemotherapy (CT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The Experimental Group participants will be submitted to the inhalation of the hedonic aroma during the chemotherapeutic treatment, this being the intervention of the study.The control group is not subject to intervention.
  Interventions: Biological: Inhalation of essential oils
- Control Group (No Intervention): The control group is not subject to intervention.

INTERVENTIONS:
Biological: Inhalation of essential oils — Intervention "Inhalation of essential oils": From the T1 (2nd Cycle CT), Experimental Group Arms will undergo the inhalation of the hedonic aroma selected by them at the time of chemotherapy (among several types of aromas). It is intended that the participant, when receiving the CT, inhales the aroma phase-in and under the investigator's observation until the end of the treatment (about two hours). The inhalation of essential oils will occur using cotton rolls impregnated with the selected oil. The control group is not subject to intervention during chemotherapy treatment.
  Arms: Experimental Group

SUMMARY:
Breast cancer is a major public health problem and is the main cancer disease in women worldwide and in Europe. In Portugal it is the most common cancer, the third cause of cancer death, following the European trend.

Breast cancer (BC) triggers a myriad of physical and psychosocial stressors with repercussions on quality of life (QoL). This study is a pioneering Randomized Controlled Trial (RCT) in Portugal, which seeks to study the impact of a hedonic aroma during chemotherapy on women with breast cancer (3, 6 and 9 weeks, and 3 months after completion of chemotherapy). To this end, participants will be randomly assigned to one of the groups. The experimental group (EG) will be exposed to chemotherapy together with a hedonic aroma, while the control group (CG) will only be exposed to chemotherapy. Both groups will be assessed on psychological morbidity, illness perception, self-efficacy for coping, executive function, cortisol levels, side-effects, beliefs about chemotherapy and QoL.

The aim of this study is to assess the impact of a hedonic aroma on the clinical, emotional and neurocognitive variables that contribute to reducing the side effects of chemotherapy and promoting QoL in women with BC.

DETAILED DESCRIPTION:
The sample is non-probabilistic, consisting of 56 participants in the control group (CG) and 56 in the experimental group (EG). According to the calculations made for RCT studies (Noordzij et al., 2010), it will take approximately a total of 100 participants (50 participants per group) to detect a 10-point difference between the groups in the result variable QoL (e.g. EORCT QLQ-C30), with a population standard deviation of 15.43, according to previous study data (Lua et al., 2015), assuming a power of 90% and a significance level of 5%.

This study contemplates four moments of evaluation: T1 (baseline: 2nd Cycle of CT but before intervention), T2 (6 weeks - 3rd Cycle), T3 (9 weeks - 4th Cycle) and T4 (3 months after the end of the CT). These moments were chosen taking into account the classes of drugs used in the CT. Each cycle has an interval of 21. This is a randomized controlled clinical trial (RCT) being single blind (the participant does not know which group he belongs to, only the investigator) and longitudinal.

Intervention procedure:

From the 2nd. Chemotherapy cycle (T1), the GC received the standard chemotherapy treatment; while the EG, in addition to the standard chemotherapy treatment, inhaled a hedonic aroma selected at the time of the chemotherapy (among three types of essential oils: bergamot, exotic verbena and geranium). The participant, as she received the CT, would inhale the aroma in a phased manner and under the supervision of the researcher, until the end of the treatment (about two hours). This intervention took place over three cycles of CT (2nd, 3rd and 4th Cycles). Inhalation was carried out using cotton rolls impregnated with the selected oil, since the more directly the odoriferous molecules are applied to the nose, the greater their impact into the organism (Schneider, 2016). However, since it was necessary that the researcher supervised the participants during the inhalation process, the number of times the researcher was in contact with participants from both groups (GC and EG) were the same: 4 times during the chemotherapy treatment to assure the participants from the EG would not have more contacts what could bias the results.

ELIGIBILITY:
Inclusion Criteria:

* women with BC in stages 0-2;
* level 0-2 on the Zubrod scale,
* without cognitive impairment,
* adjuvant chemotherapy (AQ) treatment.

Exclusion Criteria:

* Severe mental disturbance;
* olfactory impairment (≤6), evaluated before CT through the instrument smell diskettes and only in the EG participants

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2019-04-04 (Actual); Study Completion 2019-04-04 (Actual)

PRIMARY OUTCOMES:
Quality of life - The experimental group presented, in comparison to the control group, lower level of QLQ | Changes from the 2nd cycle of CT(T1) (each cycle takes, on average, 2 hours with 3-week intervals) until 4th cycle of CT, assessed up to an average 1,5 months (T3) and again in the follow up (T4) (3 months after to the end CT, an average 6 months
  Assessment instruments: the European Organization for Research and Treatment of Cancer - Quality of Life (EORTC QLQ-C30) (Aaronson et al., 1993; Pais-Ribeiro, Pinto & Santos, 2008). Interpretation of the results, the higher the value obtained, the better the total quality of life - total quality of life result, through weighting formulas carried out by the European Organization for Research and Treatment of Cancer (EORTC) (http://groups.eortc.be/qol/manuals)
Anxiety and depression - The experimental group presented, in comparison to the control group, lower anxiety and depression | Changes from the 2nd cycle of CT(T1) (each cycle takes, on average, 2 hours with 3-week intervals) until 4th cycle of CT, assessed up to an average 1,5 months (T3) and again in the follow up (T4) (3 months after to the end CT, an average 6 months
  Assessment instruments: Hospital Anxiety and Depression Scale (HADS, Pais-Ribeiro et al., 2007) comprising both anxiety and depression scales. Scores range between 0 and 42 (anxiety between 0 and 21 and depression the same), with higher results indicating higher levels of distress.

SECONDARY OUTCOMES:
Distress | Changes from the 2nd cycle of CT(T1) (each cycle takes, on average, 2 hours with 3-week intervals) until 4th cycle of CT, assessed up to an average 1,5 months (T3) and again in the follow up (T4) (3 months after to the end CT, an average 6 months
  Assessment instruments: Emotions Thermometer (TE, Mitchell, Baker-Glenn, Granger, & Symonds, 2010; Teixeira et al., 2019) consisting of five analogue-visual scales, with four domains to identify emotional complications (distress, anxiety, depression, anger) and one outcome domain (need for help). In each thermometer de scores range between 0 and 10. A high result indicates emotional distress.
Saliva cortisol | Changes from the 2nd cycle of CT(T1) (each cycle takes, on average, 2 hours with 3-week intervals) until 4th cycle of CT, assessed up to an average 1,5 months (T3) and again in the follow up (T4) (3 months after to the end CT, an average 6 months
  The collection of saliva for the evaluation of cortisol concentrations was performed using salivettes® (Starsedt). The procedure to assess salivary cortisol concentrations was implemented according to the protocol stipulated by IBL International (Cortisol Saliva ELISA, IBL International GMBH).
Subscales of the Quality of Life in Breast Cancer | Changes from the 2nd cycle of CT(T1) (each cycle takes, on average, 2 hours with 3-week intervals) until 4th cycle of CT, assessed up to an average 1,5 months (T3) and again in the follow up (T4) (3 months after to the end CT, an average 6 months
  Assessment instruments: the European Organization for Research and Treatment of Cancer - Quality of Life, Module for Breast Cancer (EORTC QLQ-BR23, Sprangers et al., 2006. In this study, only the breast symptoms (scores range between 4-16), body image (scores range between 4-16), sexual functioning (scores range between 2-8) and side effects (scores range between 7-28) subscales were used. High scores indicate higher body image, sexual functioning and breast symptoms.
Illness Perceptions | Changes from the 2nd cycle of CT(T1) (each cycle takes, on average, 2 hours with 3-week intervals) until 4th cycle of CT, assessed up to an average 1,5 months (T3) and again in the follow up (T4) (3 months after to the end CT, an average 6 months
  Assessment instruments: Illness Perception Questionnaire (IPQ-Brief, Broadbent, Petrie, Main, & Weinman, 2006; Figueiras et al., 2010). This instrument comprises 9 items that assess patients' cognitive and emotional representations of the disease. There is one item that is open-ended and asks the perceived causes of the disease (not used in the study). Scores range between 0 and 80. Higher scores indicate a more threatening illness perception.
Self-efficacy for coping | Changes from the 2nd cycle of CT(T1) (each cycle takes, on average, 2 hours with 3-week intervals) until 4th cycle of CT, assessed up to an average 1,5 months (T3) and again in the follow up (T4) (3 months after to the end CT, an average 6 months
  Assessment instruments: Cancer Behavior Inventory-Brief Version (CBI-B, Heitzmann et al., 2011). This instrument evaluates self-efficacy for coping in cancer patients through 12-item. Scores range between 12 and 108 and higher scores indicate more effective coping strategies.
Working memory | Changes from the 2nd cycle of CT(T1) (each cycle takes, on average, 2 hours with 3-week intervals) until 4th cycle of CT, assessed up to an average 1,5 months (T3) and again in the follow up (T4) (3 months after to the end CT, an average 6 months
  Assessment instruments: WAIS III Subtest - Digit Span (Wechsler, 2008). It evaluates patients' working memory in clinical practice consisting of two parts: The Digit Span Forward (scores range between 0-16 maximum) and Digit Span Backward (DSB) (scores range between 0-14 maximum). High scores indicate high immediate auditory memory and working memory.
Cognitive Flexibility | Changes from the 2nd cycle of CT(T1) (each cycle takes, on average, 2 hours with 3-week intervals) until 4th cycle of CT, assessed up to an average 1,5 months (T3) and again in the follow up (T4) (3 months after to the end CT, an average 6 months
  Assessment instruments: Trail Making Test (TMT, Partington & Leiter, 1949; Cavaco et al., 2013). This instrument is composed of part A, which evaluates attention, visual tracking and speed of graphomotor coordination and information processing; and Part B evaluates Part A functions and the ability to switch between a set of stimuli. Lower raw indices and higher adjusted scores correspond to better cognitive performance.
Beliefs about chemotherapy | Changes from the 2nd cycle of chemotherapy (T1) (each cycle takes, on average, 2 hours with 3-week intervals between each cycle) until the date of 4th cycle of CT, assessed up to an average 1,5 months (T3)
  Assessment instruments: Beliefs about chemotherapy (BMQ, Horne, Weinman, & Hankins, 1997; Pereira, Pedras, & Machado, 2013). This instrument is composed of 18 items and comprises two sections: BMQ - Specific and BMQ-General. In this study, only the specific section was used regarding chemotherapy. The BMQ - Specific section incorporates two sub-scales of five items each: Specific Needs and Specific Concerns related to the dangers of dependence and toxicity and concerns regarding long-term side effects, respectively. The total on the Specific Needs Scale ranges from 5 to 25 and on the Specific Concerns Scale from 5 to 25. Higher scores in each subscale indicate stronger beliefs regarding the need of treatment and regarding concerns towards the treatment, respectively.

OTHER OUTCOMES:
Sociodemographic and Clinical Data | Time Frame: before chemotherapy (CT) treatment
  Assessment instruments: This instrument was developed specifically for this study, and included 11 items to assess sociodemographic variables (age, marital status, education, and occupation) and clinical variables (type of surgery, disease stage, number of planned cycles, tumor grade, sentinel lymph node, molecular markers and take hormone therapy).
ECOG Performance Status (Oken et al., 1982) | Time Frame: before CT for inclusion criteria
  The Zubrod scale evaluates patients' performance status, where 0 refers to fully functional and asymptomatic and 5 to dead. It was used for inclusion criteria (West & Jin, 2015).
Smell Diskettes (Simmen, Briner & Hess, 1999). | Time Frame: before CT for inclusion criteria
  This test consists of eight reusable diskettes containing different odors. It is a test that aims to evaluate the olfactory function. According to the results, a score between 7 and 8 corresponds to a normal olfactory function and ≥6 presents a compromised olfactory function (as for example with a hyposmia or anosmia).
Short Assessment of Health Literacy (SAHL, Lee et al., 2010; Apolinario et al., 2012). | Time Frame: before CT for inclusion criteria
  This instrument assesses the degree of health literacy through the recognition of medical words, associating them with other words of similar meaning. Higher scores indicate a higher level of health literacy. A cutoff point of <14 has been assumed to distinguish between adequate and inadequate literacy (Apolinario et al., 2012).

CONTACTS AND LOCATIONS:
Overall Officials: Marta Pereira, Master, Principal Investigator — University of Minho
Locations (1):
- António Fradão, Viana do Castelo, Estrada de Santa Luzia, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Apolinario D, Braga Rde C, Magaldi RM, Busse AL, Campora F, Brucki S, Lee SY. Short Assessment of Health Literacy for Portuguese-speaking Adults. Rev Saude Publica. 2012 Aug;46(4):702-11. doi: 10.1590/s0034-89102012005000047. Epub 2012 Jul 10. PMID 22782124
- [Background] Broadbent E, Petrie KJ, Main J, Weinman J. The brief illness perception questionnaire. J Psychosom Res. 2006 Jun;60(6):631-7. doi: 10.1016/j.jpsychores.2005.10.020. PMID 16731240
- [Background] Cavaco S, Goncalves A, Pinto C, Almeida E, Gomes F, Moreira I, Fernandes J, Teixeira-Pinto A. Trail Making Test: regression-based norms for the Portuguese population. Arch Clin Neuropsychol. 2013 Mar;28(2):189-98. doi: 10.1093/arclin/acs115. Epub 2013 Jan 7. PMID 23299183
- [Background] Figueiras M, Marcelino DS, Claudino A, Cortes MA, Maroco J, Weinman J. Patients' illness schemata of hypertension: the role of beliefs for the choice of treatment. Psychol Health. 2010 Apr;25(4):507-17. doi: 10.1080/08870440802578961. PMID 20204931
- [Background] Heitzmann CA, Merluzzi TV, Jean-Pierre P, Roscoe JA, Kirsh KL, Passik SD. Assessing self-efficacy for coping with cancer: development and psychometric analysis of the brief version of the Cancer Behavior Inventory (CBI-B). Psychooncology. 2011 Mar;20(3):302-12. doi: 10.1002/pon.1735. PMID 20878830
- [Background] Lee SY, Stucky BD, Lee JY, Rozier RG, Bender DE. Short Assessment of Health Literacy-Spanish and English: a comparable test of health literacy for Spanish and English speakers. Health Serv Res. 2010 Aug;45(4):1105-20. doi: 10.1111/j.1475-6773.2010.01119.x. Epub 2010 May 24. PMID 20500222
- [Background] Mitchell AJ, Baker-Glenn EA, Granger L, Symonds P. Can the Distress Thermometer be improved by additional mood domains? Part I. Initial validation of the Emotion Thermometers tool. Psychooncology. 2010 Feb;19(2):125-33. doi: 10.1002/pon.1523. PMID 19296462
- [Background] Noordzij M, Tripepi G, Dekker FW, Zoccali C, Tanck MW, Jager KJ. Sample size calculations: basic principles and common pitfalls. Nephrol Dial Transplant. 2010 May;25(5):1388-93. doi: 10.1093/ndt/gfp732. Epub 2010 Jan 12. PMID 20067907
- [Background] Horne R, Weinman J, Hankins M. The beliefs about medicines questionnaire: the development and evaluation of a new method for assessing the cognitive representation of medication. Psychology and health. 1999; 14(1): 1-24.
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Background] Pais-Ribeiro JL, Pinto C, Santos C. Validation study of the Portuguese version of the QLC-C30-V. 3. Psicologia, Saúde & Doenças. (2008; 9(1): 89-102.
- [Background] Pais-Ribeiro J, Silva I, Ferreira T, Martins A, Meneses R, Baltar M. Validation study of a Portuguese version of the Hospital Anxiety and Depression Scale. Psychol Health Med. 2007 Mar;12(2):225-35; quiz 235-7. doi: 10.1080/13548500500524088. English, Portuguese. PMID 17365902
- [Background] Partington JE, Leiter RG. Partington's pathway test. Psychological Service Center Bulletin. 1949; 9-20.
- [Background] Schneider R. There Is Something in the Air: Testing the Efficacy of a new Olfactory Stress Relief Method (AromaStick(R)). Stress Health. 2016 Oct;32(4):411-426. doi: 10.1002/smi.2636. Epub 2015 Mar 18. PMID 25787105
- [Background] Simmen D, Briner HR, Hess K. [Screening of olfaction with smell diskettes]. Laryngorhinootologie. 1999 Mar;78(3):125-30. doi: 10.1055/s-2007-996844. German. PMID 10226979
- [Background] Sprangers MA, Groenvold M, Arraras JI, Franklin J, te Velde A, Muller M, Franzini L, Williams A, de Haes HC, Hopwood P, Cull A, Aaronson NK. The European Organization for Research and Treatment of Cancer breast cancer-specific quality-of-life questionnaire module: first results from a three-country field study. J Clin Oncol. 1996 Oct;14(10):2756-68. doi: 10.1200/JCO.1996.14.10.2756. PMID 8874337
- [Background] Teixeira RJ, Machado JC, Faria S, Remondes-Costa S, Brandao T, Branco M, Moreira S, Pereira MG. Brief emotional screening in oncology: Specificity and sensitivity of the emotion thermometers in the Portuguese cancer population. Palliat Support Care. 2020 Feb;18(1):39-46. doi: 10.1017/S1478951519000208. PMID 31164179
- [Background] Wechsler D. Escala de Inteligência de Wechsler para Adultos-Terceira Edição [Wechsler Adult Intelligence Scale-Third Edition] (WAIS-III). Lisboa: Cegoc. 2008
- [Background] West HJ, Jin JO. JAMA Oncology Patient Page. Performance Status in Patients With Cancer. JAMA Oncol. 2015 Oct;1(7):998. doi: 10.1001/jamaoncol.2015.3113. No abstract available. PMID 26335750
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Pereira MG, Pedras S, Machado JC. Validation of the questionnaire of beliefs towards medicines in type 2 diabetic patients. Psicologia: Teoria e Pesquisa. 2013; 29: 229-236.
- [Derived] Pereira M, Moreira CS, Izdebski P, Dias ACP, Nogueira-Silva C, Pereira MG. How Does Hedonic Aroma Impact Long-Term Anxiety, Depression, and Quality of Life in Women with Breast Cancer? A Cross-Lagged Panel Model Analysis. Int J Environ Res Public Health. 2022 Jul 28;19(15):9260. doi: 10.3390/ijerph19159260. PMID 35954612